CLINICAL TRIAL: NCT00390468
Title: A Phase II Study of Tandutinib (MLN518) in Androgen-Independent Prostate Cancer With Bone Metastases
Brief Title: Tandutinib in Treating Patients With Progressive Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02865; P30CA016672 (NIH); MDA-2005-0717 (Other: UT MD Anderson Cancer Center); NCI-7409; CDR0000504104 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Cancer; Pain; Prostate Cancer
Keywords: Tandutinib; MLN518; CT53518; pain; adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; bone metastases; hormone-based castration
MeSH Terms: conditions — Neoplasm Metastasis; Pain; Prostatic Neoplasms | interventions — tandutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tandutinib (MLN518) (Experimental): 500 mg twice daily, a small-molecule inhibitor of the type III receptor tyrosine kinases. Tandutinib (MLN518) previously known as CT53518.
  Interventions: Drug: Tandutinib

INTERVENTIONS:
Drug: Tandutinib — 500 mg twice daily every day with doses taken approximately 12 hours apart, 28 day cycle.
  Other Names: CT53518

SUMMARY:
RATIONALE: Tandutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well tandutinib works in treating patients with progressive prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with progressive androgen-independent prostate cancer with bone metastases treated with tandutinib.

Secondary

* Determine the prostate-specific antigen (PSA) decline rate by 50% (PSA response), using the PSA Working Group Criteria, in patients treated with this regimen .
* Evaluate modulation of bone pain and bone markers in patients treated with this regimen.
* Determine the objective tumor response by RECIST (Response Evaluation Criteria In Solid Tumors) criteria in patients treated with this regimen.
* Determine the qualitative and quantitative toxicity of this regimen in these patients.

OUTLINE: Patients receive oral tandutinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Bone pain is assessed at baseline, on day 1 of course 3, and at disease progression.

After completion of study treatment, patients are followed for 4 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate.
2. Patients must have radiological evidence of bone metastases.
3. Patients must have a castrate level of testosterone (</= 50ng/ml). For patients who are medically castrated, luteinizing hormone releasing hormone analog must continue to maintain testicular suppression.
4. Patients must have evidence of progressive disease (e.g. progressive bone pain from bone metastases, increasing bidimensional disease on clinical examination or X-rays or appearance of new lesions on bone radiographs). Alternatively, for patients without such evidence of progression, PSA-progression is defined by 2 consecutive rises in prostate-specific antigen (PSA), each an absolute change of at least 1ng/ml, measured at least 2 weeks apart.
5. A minimum PSA >/= 5ng/ml is required.
6. Patients on anti-androgens should be discontinued from such therapy for at least 4 weeks (for bicalutamide for at least 6 weeks), unless there is interim evidence of progression as defined in Inclusion #4.
7. Patients must have had one prior taxane-based regimen but no prior known PDGFR, platelet-derived growth factor receptor, inhibitor (e.g. imatinib, SU11248, BAY43-9006) therapy is permitted.
8. Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of TANDUTINIB in patients < 18 years of age, children are excluded from this study.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
10. Patients must have adequate organ and marrow function as follows: leukocytes >/= 3,000/mcL; absolute neutrophil count >/= 1,500/mcL; platelets >/= 100,000/mcL; total bilirubin within normal institutional limits; aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </= 2.5 times institutional upper limit of normal; creatinine within normal institutional limits OR creatinine clearance >/= 40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
11. The effects of TANDUTINIB on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because receptor tyrosine kinase inhibitors are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control, or abstinence) prior to study entry and for 3 months after completion of study therapy.
12. Ability to understand and the willingness to sign a written informed consent document.
13. Men of all races and ethnic groups are eligible for this trial. This is a study in prostate cancer and is therefore not applicable to women.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from dose-limiting adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents or hormonal therapy besides that used to maintain medical castration. Glucocorticoid therapy for intercurrent medical illnesses such as asthma, Chronic Obstructive Pulmonary Disease (COPD) or rheumatoid arthritis flare will be allowed.
3. Patients may not be co-medicated with an agent that causes QTc prolongation.
4. Patients with a mean QTc >500msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome are ineligible.
5. Left ventricular ejection fraction (LVEF) <40%.
6. Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
7. Ongoing vomiting, or nausea >/= Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0). If nausea, or vomiting is controlled with therapy (and therefore not Grade 2) such patients may be enrolled.
8. Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow pills or absorb oral medications are excluded.
9. History of chronic liver disease.
10. Known or suspected primary muscular or neuromuscular disease (e.g., muscular dystrophy, myasthenia gravis).
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to tandutinib. Patients who develop an acneiform/maculopustular rash while taking either gefitinib or erlotinib should not be prevented from receiving tandutinib unless the rash is considered an allergic reaction (angioedema/urticaria) or Stevens-Johnson syndrome.
12. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections defined as requiring IV antibiotics on Day 1 of treatment or psychiatric illness/social situations that would limit compliance with study requirements.
14. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with TANDUTINIB. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Result] Mathew P, Tannir N, Tu SM, Wen S, Guo CC, Marcott V, Bekele BN, Pagliaro L. Accelerated disease progression in prostate cancer and bone metastases with platelet-derived growth factor receptor inhibition: observations with tandutinib. Cancer Chemother Pharmacol. 2011 Oct;68(4):889-96. doi: 10.1007/s00280-011-1567-2. Epub 2011 Feb 3. PMID 21290244
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at UT MD Anderson Cancer Medical Clinic from October 24, 2006 to January 8, 2008.
Pre-assignment Details: Participants must have had at least one prior taxane based regimen but no prior known Platelet Derived Growth Factor Receptor (PDGFR) inhibitor therapy was permitted.
Groups:
- Tandutinib (MLN518): 500 mg twice daily, a small-molecule inhibitor of the type III receptor tyrosine kinases
Period: Overall Study
Arm/Group | Tandutinib (MLN518)
Started | 18
Completed | 15
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tandutinib (MLN518)
Number analyzed (Participants) | 18
Age, Customized [Median (Full Range); unit: years] | 66 [47 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: 8-week Freedom-From-Progression (FFP)
Description: Simon 2 stage design for freedom from progression at 8 weeks where time-to-progression defined as time of initiation of therapy to first determination of progression of disease by clinical, radiological or serological criteria: Frequency of p-PDGFR (phosphorylated platelet-derived growth factor receptor) expression in bone marrow biopsy specimens, prostate-specific antigen (PSA) declines by 50% sustained for 4 weeks, measurable disease outcomes by RECIST (Response Evaluation Criteria In Solid Tumors) criteria, and quantitative/qualitative toxicities assessed.
Time Frame: 8 weeks; repeat assessments performed every 8 weeks after criteria for response first met.
Population: Analysis was per protocol; Of 18 participants, only 15 were evaluable for efficacy.
Measure: Number; unit: participants
Arm/Group | Tandutinib (MLN518)
Number analyzed (Participants) | 18
participants
  Participants Progression Free at 8 Weeks | 2 [3 to 40]
  Evaluable Participants at 8 Weeks | 15

ADVERSE EVENTS:
Time Frame: 14 months
Description: The following scale grades adverse events by common features: Grade 1 = Mild Severity; Grade 2 = Moderate Severity; Grade 3 = Serious Severity.
Arm/Group | Tandutinib (MLN518)
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandutinib (MLN518) (N=15)
Cranial Nerve III (Nervous system disorders) | 1 (1)
platelet count low (Blood and lymphatic system disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
infection with normal ANC (Immune system disorders) | 1 (1) — Absolute neutrophil count (ANC)
pulmonary obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hemmorhage GU urinary NOS (Renal and urinary disorders) | 1 (1) — GU (Genitourinary) urinary nitric oxide synthase (NOS)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandutinib (MLN518) (N=15)
nausea (Gastrointestinal disorders) | 15 (22) — grade 1 & 2
vomiting (Gastrointestinal disorders) | 15 (16) — grade 1 & 2
fatigue (General disorders) | 15 (23) — grade 1, 2, & 3
anemia (Blood and lymphatic system disorders) | 15 (26) — grade 1, 2, and 3

LIMITATIONS AND CAVEATS:
The study was closed to further accrual per design specifications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less